CLINICAL TRIAL: NCT07093866
Title: Efficacy and Safety of Disitamab Vedotin Plus Abiraterone for Metastatic Castration-Resistant Prostate Cancer：a Phase II Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Nanjing University (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-125
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: mCRPC
Keywords: mCRPC
MeSH Terms: interventions — disitamab vedotin; RC48 antibody; abiraterone; Prednisone

STUDY DESIGN:
Intervention Model Description: Experimental regimen: Disitamab vedotin +Abiraterone +Prednisone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): mCRPC subjects with IHC 1+/IHC 2+/IHC3+ are administered Disitamab Vedotin combined with Abiraterone
  Interventions: Drug: Disitamab Vedotin (RC48); Drug: Abiraterone + prednisone

INTERVENTIONS:
Drug: Disitamab Vedotin (RC48) — Disitamab Vedotin 2mg/kg is administered intravenously once every 2 weeks (1 cycle)
Drug: Abiraterone + prednisone — Abiraterone 1000mg is administered orally once a day，and prednisone 5mg is administered orally twice a day.

SUMMARY:
This is an open-label，prospective，single-arm，phase 2 trial aims to evaluate the efficacy and safety of disitamab vedotin combined with abiraterone in patients with metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients are able to understand and voluntarily sign the informed consent form (ICF); judged by the investigator to be capable of complying with the protocol.
* Male patients of ≥18 years or older at the time of ICF signature.
* Patients with ECOG performance status 0-1.
* Patients with an expected survival of 3months or more.
* Patients who are histologically or cytologically confirmed prostatic adenocarcinoma with HER2 expression (IHC 1+, 2+ or 3+) in archival or fresh tumour tissue.
* Patients with documented castration-resistant prostate cancer (CRPC): serum testosterone <1.73 nmol/L (50 ng/dL) at screening; patients on medical castration must continue LHRH agonist/antagonist therapy throughout the study.
* Patients with evidence of metastatic disease by bone scan (bone lesions) and/or CT/MRI (soft-tissue lesions).
* Patients with adequate organ function as defined below:

  * Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L
  * Platelet count (PLT) ≥100 × 10⁹/L
  * Hemoglobin (Hb) ≥100 g/L
  * Total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN); ≤2 × ULN if liver metastases present
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 × ULN; ≤2 × ULN if liver metastases present
  * Serum creatinine (Cr) ≤1.5 × ULN or calculated creatinine clearance (CrCl) ≥60 mL/min (Cockcroft-Gault formula; calculate only if Cr >1.5 × ULN)
  * Urinalysis protein <2+; if ≥2+, 24-h urine protein must be <1 g or urine protein/creatinine ratio <0.5
  * For patients not on anticoagulation: INR and aPTT ≤1.5 × ULN; patients on stable-dose anticoagulation are eligible
  * Left ventricular ejection fraction (LVEF) ≥50% or ≥local lower limit of normal (LLN), whichever is lower
  * QTcF interval <470 ms
* Male patients with partners of child-bearing potential must use a medically acceptable contraceptive method from the first study dose until 3 months after the last dose.

Exclusion Criteria:

* Patients who are known hypersensitivity to any component of disitamab vedotin or abiraterone.
* Patients with other malignancies within 3 years before screening, except early-stage malignancies considered clinically cured (carcinoma in situ or stage I tumors), e.g., basal-cell or squamous-cell skin carcinoma or superficial bladder cancer.
* Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with treated brain metastases may enroll if lesions have been stable for ≥1 month, there is no evidence of new or enlarging CNS disease, and systemic corticosteroids have been discontinued ≥3 days before the first study dose.
* Patients who are clinically significant pericardial effusion, or pleural/peritoneal/pelvic effusions that are poorly controlled or require drainage within 2 weeks before the first dose.
* Patients with major surgical intervention (any grade 3 or 4 procedure per the 2009 Chinese Regulation on Clinical Application of Medical Technologies) within 4 weeks before the first dose, or incomplete post-operative recovery that, in the investigator's judgment, poses a risk to trial participation.
* Patients who are prior PSMA-targeted therapy.
* Patients within 4 weeks (6 weeks for nitrosoureas or mitomycin C) before the first dose: any antineoplastic chemotherapy (except castration therapy), radiotherapy (>1 week of local palliative radiotherapy permitted), endocrine therapy (estrogens or anti-androgens; bicalutamide or nilutamide require 6-week washout), targeted therapy, immunotherapy, or participation in another interventional clinical trial (observational studies or post-trial follow-up are allowed).

  * Patients with stable-dose denosumab or bisphosphonates for bone metastases are permitted.
  * mCRPC patients must not have used PSA-lowering herbal agents (e.g., saw palmetto) or systemic corticosteroids (except short courses for allergy prophylaxis/treatment) within 4 weeks before the first dose, nor plan to use such agents during the study.
* Patients with use of antineoplastic traditional Chinese medicine (TCM) prescriptions or proprietary TCM within 1 week, or receipt of blood transfusion/blood products, hematopoietic growth factors, or other agents to correct blood cell counts within 2 weeks before first study dose.
* Patients with toxicities from prior antineoplastic therapy that have not resolved to baseline, CTCAE v5.0 grade 0-1 (except alopecia and pigmentation), or to the levels specified in the inclusion/exclusion criteria; unhealed wounds. Irreversible toxicities not expected to worsen with study drug (e.g., hearing loss) are permitted.
* Patients with unexplained fever >38.5 °C (tumor-related fever may be allowed per investigator judgment); active or persistent infection; HIV antibody positive; HBsAg positive with HBV DNA > site ULN, or HBsAg-negative/HBcAb-positive with HBV DNA > site ULN after treatment; HCV antibody positive with HCV RNA > site ULN; active syphilis (except adequately treated, cured, or stable syphilis).
* NYHA class III/IV congestive heart failure; uncontrolled arrhythmia despite treatment/intervention; risk of QT prolongation or use of drugs known to prolong QT; refractory hypertension (hypertension controlled to <140/90 mmHg on medication is allowed).
* Patients with clinically significant vascular events within 6 months before first dose, including acute arterial/venous thromboembolism, thrombotic arteritis, thrombophlebitis, acute pulmonary embolism, acute coronary syndrome (MI, unstable angina, etc.), acute cerebrovascular events, or disseminated intravascular coagulation.
* Patients with tumor metastases with clear invasion of major arteries posing a high bleeding risk.
* Patients with interstitial pneumonitis, pulmonary fibrosis, or other severe pulmonary disease requiring treatment; hemoptysis >2.5 mL per episode within 3 weeks before first dose.
* Patients with active gastro-intestinal ulcer, perforation, and/or fistula requiring treatment within 6 months; GI bleeding (hematemesis, melena, or hematochezia) within 3 months without endoscopic/colonoscopic evidence of complete healing.
* Patients with uncontrolled concurrent disease >CTCAE v5.0 grade 2 (e.g., diabetes).

Uncontrolled concurrent disease >CTCAE v5.0 grade 2 (e.g., diabetes).

* Patients with CTCAE v5.0 grade >2 peripheral neuropathy, prior epilepsy, psychiatric disorders; history of drug abuse within 6 months or alcohol abuse within 3 months (alcohol abuse defined as >14 units/week: 1 unit = 285 mL beer, 25 mL spirits, or 80 mL wine).
* Patients with autoimmune disease, immunodeficiency, or organ transplantation.
* Patients with any condition, therapy, or laboratory abnormality that, in the investigator's opinion, could confound results, interfere with trial participation, or be not in the subject's best interest.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
PSA 50 | baseline up to 24 weeks
  Proportion of patients with a ≥50 % prostate-specific antigen (PSA) reduction from baseline at Week 12, confirmed by a repeat assessment at least 3 weeks later.

SECONDARY OUTCOMES:
PSA 30 | baseline up to 24 weeks
  Proportion of patients with a ≥30 % prostate-specific antigen (PSA) reduction from baseline at Week 12, confirmed by a repeat assessment at least 3 weeks later.
PSA 90 | baseline up to 24 weeks
  Proportion of patients with a ≥90 % prostate-specific antigen (PSA) reduction from baseline at Week 12, confirmed by a repeat assessment at least 3 weeks later.
Radiographic Progression-Free Survival（rPFS） | From baseline until radiographic progression or death from any cause, whichever comes first. assessed up to 36 months
  Time from the first day of study drug administration to the earlier of radiographic progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu 210000, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No